CLINICAL TRIAL: NCT06680089
Title: A Study of the Clinical Application of [18F]RCCB6 PET/ CT Imaging in the Diagnosis of Kidney Cancer
Brief Title: CD70-targeted immunoPET Imaging of Kidney Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LY2024-138-A
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Urologic Neoplasms; Urogenital Neoplasms; Kidney Neoplasms; Neoplasms
Keywords: The cluster of differentiation (CD70); Kidney tumor; Clear cell renal cell carcinoma; ImmunoPET
MeSH Terms: conditions — Urologic Neoplasms; Urogenital Neoplasms; Kidney Neoplasms; Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD70-targeted immunoPET imaging (Experimental): Enrolled patients will undergo a CD70-targeted immunoPET/CT scanning.
  Interventions: Drug: [18F]RCCB6

INTERVENTIONS:
Drug: [18F]RCCB6 — Enrolled patients will receive 0.05-0.1mCi/kg of [18F]RCCB6. ImmunoPET/CT imaging will be acquired 1 hour after [18F]RCCB6 injection.
  Other Names: [18F]F-RESCA-RCCB6

SUMMARY:
The aim of this study is to establish and optimize the [18F]RCCB6 PET/CT imaging method, and its physiological and pathological distribution characteristics, on the basis of which the diagnostic efficacy of the above imaging agent in renal cancer (especially clear cell renal cell carcinoma) wil be evaluated.

DETAILED DESCRIPTION:
Histologically confirmed diagnosis of kidney cancer (especially clear cell renal cell carcinoma and papillary renal cell carcinoma) or suspected kidney cancer by diagnostic imaging will be included. Especially patients with suspected metastases or routine follow-up or surveillance or suitable for systemic treatments (e.g., combined immunotherapy and targeted therapies) will undergo [18F]RCCB6 immunoPET/CT scans. Enrolled patients will undergo whole-body [18F]RCCB6 immunoPET/CT scans at 1 hour after tracer injection(0.05-0.1 mCi/kg). Uptake of [18F]RCCB6 in tumor and normal organs/tissues will be scored visually and quantitatively. Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to evaluate the diagnostic efficacy. Furthermore, we will compare the diagnostic rates of [18F]RCCB6 immunoPET/CT with those of conventional imaging examinations, such as CT, MRI, and 18F-FDG PET/CT, etc.The correlation between lesion uptake and protein expression level determined by immunohistochemistry staining will be further analyzed. Further explore the value of [18F]RCCB6 in treatment decision-making（staging, surveillance, and restaging） for kidney cancer.We will conduct an interim assessment when more than half of the patients have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 year-old and of either sex；
2. Histologically confirmed diagnosis of kidney cancer (especially clear cell renal cell carcinoma and papillary renal cell carcinoma) or suspected kidney cancer by diagnostic imaging;
3. Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.

Exclusion Criteria:

1. Pregnancy；
2. Severe hepatic and renal insufficiency;
3. History of serious surgery in the last month;
4. Allergic to antibody or single-domain antibody radiopharmaceuticals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of [18F]RCCB6 | 1 day from injection of the tracer
  Measurement of the overall biodistribution of [18F]RCCB6 in normal tissues and organs.
Standardized uptake value (SUV) | 1 day from injection of the tracer
  Standardized uptake value (SUV) of [18F]RCCB6 in the included subjects' primary and/or metastatic lesions.
The correlation between CD70 expression and [18F]RCCB6 uptake value | 60 days
  The Standardized uptake value (SUV) of [18F]RCCB6 will be calculated, and the correlation between pathological results and tumor uptake of [18F]RCCB6 will be analyzed.
Diagnostic value of [18F]RCCB6 PET in patients with ccRCC | 30 days
  We will calculate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy of [18F]RCCB6 PET/CT in patients with ccRCC. We will also compare the diagnostic value of [18F]RCCB6 with that of traditional imaging tracers (e.g., 18F-FDG) and imaging modalities (e.g., CT and MRI). All the above goals will be achieved by analyzing the static/dynamic [18F]RCCB6 PET/CT imaging data. Systematic evaluation of these parameters will elucidate the pharmacokinetics, pharmacodynamics, and, more importantly, the clinical value of [18F]RCCB6 PET/CT for patients with ccRCC.
To explore the diagnostic performance of [18F]RCCB6 PET with that of conventional imaging and [18F]FDG PET | 6 months
  Using pathological or follow-up imaging data as the gold standard, explore the diagnostic performance of [18F]RCCB6 PET compared to conventional imaging and [18F]FDG PET.

SECONDARY OUTCOMES:
[18F]RCCB6 PET/CT in changing clinical decision-making for ccRCC patients | 3-6 months
  After analyzing the imaging parameters and diagnostic/predictive value of [18F]RCCB6 PET/CT, we will also investigate how clinical use of [18F]RCCB6 PET/CT changes clinical decision-making for ccRCC patients. Joint efforts from nuclear medicine physicians, urologists, oncologists, and pathologists will draw solid conclusions from the imaging and clinical information.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhai, Ph.D. & M.D., Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University; Weijun Wei, Ph.D. & M.D., Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China